CLINICAL TRIAL: NCT05544669
Title: Study of Calcium-phosphate Complications Induced by the Administration of IV Iron Supplementation in Patients With Rendu-Osler Disease
Brief Title: Calcium-phosphate Complications Induced by IV Iron Supplementation in Patients With Rendu-Osler Disease
Acronym: OS-LERETRO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8696
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Rendu Osler Disease
Keywords: Rendu-Osler disease; Hypophosphatemia; Injectable iron; Osteomalacia; Carbohydrates; Iron deficiency
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Hypophosphatemia; Osteomalacia; Iron Deficiencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypophosphatemia induced by treatments with injectable iron is a frequent side effect already reported during marketing. Situations of osteomalacia secondary to these hypophosphatemias are rarer and reported in the form of case reports in the literature. Hypophosphatemia in this context is attributed to an excess of FGF-23 (defect of degradation linked to carbohydrates in martial preparations) with renal leakage of phosphate.

Rendu-Osler disease (ROM) is an autosomal dominant genetic disease, favoring the formation of vascular malformations, including nasal and digestive telangiectasias causing repeated bleeding, even hemorrhages. Iron deficiency is frequent and profound there, and oral martial treatments are often insufficient to compensate for these losses. Regular iron infusions, to avoid transfusions, are often necessary.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥ 18 years old)
* suffering from Rendu-Osler disease and receiving IV iron supplementation
* Subject not objecting, after information, to the reuse of their data for scientific research purposes

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject under safeguard of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject (≥ 18 years old) suffering from Rendu-Osler disease and receiving IV iron supplementation
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a bone crack and/or fracture | Files analysed retrospectively from January 01, 2018 to December 31, 2022 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine interne - CHU de Strasbourg - France, Strasbourg, France